CLINICAL TRIAL: NCT04372654
Title: Pilot Study Evaluating the Safety of Electroducer Sleeve Medical Device for Temporary Cardiac Stimulation During Percutaneous Cardiovascular Interventions, in All Kind of Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Electroducer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Electroducer study
Record Dates: First submitted 2020-04-28; First posted 2020-05-04 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2020-10

CONDITIONS: Coronary Disease; Valve Heart Disease; Pacemaker DDD
MeSH Terms: conditions — Coronary Disease; Heart Valve Diseases

STUDY DESIGN:
Intervention Model Description: Pilot, prospective, multicenter, non-comparative study in 60 patients with a percutaneous cardiovascular intervention indication which requires temporary cardiac stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radial group (Experimental): Use of Electroducer Sleeve on radial route
  Interventions: Device: Electroducer Sleeve
- femoral group (Experimental): Use of Electroducer Sleeve on femoral route
  Interventions: Device: Electroducer Sleeve

INTERVENTIONS:
Device: Electroducer Sleeve — The device's safety will be assessed at the radial and femoral puncture site

SUMMARY:
During percutaneous cardiovascular intervention, temporary cardiac stimulation may be required. Usually this stimulation is generated via a temporary pacing catheter. In order to reduce the complexity of the procedure, a new stimulation strategy has been developed: the "Direct Wire Pacing technique".In this approach, the cardiac stimulation is provided via the guidewire connected to an external pacemaker.

Previous study demonstrated the superiority of the new technique compared to the former. However this technique is likely to generate electrical pain, risk of bleeding for the patient and risk of blood exposure accident for the operators. This is why the medical device ELECTRODUCER SLEEVE has been developed. This device integrates a pacing function to the introducer and the guidewire used. The "Direct Wire Pacing technique" is simplified, secured and more reproducible.

DETAILED DESCRIPTION:
During percutaneous cardiovascular interventions such as Transcatheter Heart Valve or coronary intervention, temporary cardiac stimulation may be required. Usually this stimulation is generated via a temporary pacing catheter in the right ventricle. This procedure requires an additional venous access and the insertion of the stimulation catheter, which are both likely to generate complications. In order to reduce the complexity and increase the safety of the procedure, a new stimulation strategy has been developed: the "Direct Wire Pacing technique". In this approach, the specific venous access and the implantation of a stimulation catheter are avoided. The cardiac stimulation is provided via the guidewire inserted into the left ventricle or into the coronary arteries. This guidewire is connected to an external Pacemaker using an alligator clamp (Cathode). The Pacemaker anode is also connected using a clamp attached to a needle piercing the subcutaneous tissue, obtaining a closed electrical circuit. This technique was validated during previous studies in the TAVI context through two registries and one randomized controlled trial. This study demonstrated the superiority of the new technique by showing a reduction of the procedural duration, radiation exposure and costs; with similar efficacy and safety. However the subcutaneous needle insertion is likely to generate electrical pain, risk of bleeding for the patient and risk of blood exposure accident for the operators. This subcutaneous anode increases the stimulation threshold (mA) which can cause stimulation failures. Moreover, several technical difficulties preclude general adoption by the scientific community. This is why the medical device ELECTRODUCER SLEEVE has been developed. This device integrates a pacing function to the introducer and the guidewire used during percutaneous cardiovascular interventions. The guidewire then behaves like an intra-cardiac cathode. Thanks to the device, the complex manipulation of needles and clamps during the intervention are avoided as well as pole inversions. The "Direct Wire Pacing technique" used during the coronary and structural interventions is thus simplified, secured and more reproducible.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Patients with a percutaneous cardiovascular intervention indication, requiring temporary cardiac stimulation
* Procedure carried out with a 6Fr TERUMO introducer ≥ 65 mm
* Procedure performed by femoral or radial routes
* Patients able to understand and provide informed consent
* Patients able to perform the planned follow-up visit one month after the procedure.

Exclusion Criteria:

* Patients requiring a definitive PM
* Pregnant or breastfeeding woman
* Patiens under judicial protection, tutorship or curatorship
* Negative Allen test or absence of radial pulse in the artery or vein used for intervention
* Patient participating in another interventional clinical trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
To assess the peri procedural safety of ELECTRODUCER SLEEVE device used for temporary cardiac pacing during percutaneous cardiovascular interventions, by radial and femoral routes of access. | during intervention
  The device safety is assessed through the occurrence of bleeding complications at the access site where the ELECTRODUCER SLEEVE was used, including: Hematoma formation (EASY Classification) and Access-site Bleeding (BARC classification).

SECONDARY OUTCOMES:
To evaluate the occurrence of Radial Artery Occlusion | at discharge and 1 month
  RAO evaluated by a radial artery Doppler and by a reverse Allen test
To evaluate the occurrence of allergic or adverse tissue reactions | at discharge and 1 month
  Outcome evaluated through the clinical examination of the puncture site.
To establish the efficacy of the ELECTRODUCER SLEEVE device | during intervention
  Outcome evaluated through the capture in the surface electrocardiogram : each spike delivered on the guidewire is follow by its hemodynamic effect.
To evaluate the performance of the ELECTRODUCER SLEEVE device | during intervention
  Performance evaluated through the stimulation threshold (mA) measured with the external pacemaker
To evaluate the impact of the ELECTRODUCER SLEEVE use on the TAVI procedure duration. | during intervention
  Procedure duration is defined between the first vascular puncture and the last introducer removal and compared to the EASY TAVI study data
To evaluate the patient comfort with ELECTRODUCER SLEEVE use | during intervention
  Confort evaluated using the "Echelle Visuelle Analogique de la douleur" from 0 to 10: 0 being the absence of pain and 10 being unbearable pain.
To assess the user's overall impression of the ELECTRODUCER SLEEVE device and use. | during intervention
  Outcome evaluated by a satisfaction questionnaire developed by Electroducer, composed of four questions and a free comment section.

CONTACTS AND LOCATIONS:
Locations (1):
- GHMG, Grenoble, France

IPD SHARING:
Plan to Share IPD: No